CLINICAL TRIAL: NCT01209468
Title: A Randomized Clinical Trial of the Treatment of Obstructive Sleep Apnoea Using Oral Appliances
Brief Title: Treatment of Sleep Apnea With Oral Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Colman McGrath, Faculty of Dentistry, HKU
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral appliance 2 (Active Comparator): Patients in treatment arm/group B will have a customized twinblock OA constructed for them individually. They will undergo an appliance acclimatization period of 4-5 weeks. Three months after baseline assessments - T1 (6 weeks of 'active' treatment), physiological measurements will be evaluated, clinical oral examinations conducted, quality of life and compliance assessed. Following this, a customized monobloc OA will be constructed for subjects individually and they will acclimatize to it for 4-5 weeks (so that the mandible is protruded to the maximum position they feel comfortable with when the appliance is worn). Prior to the active treatment phase, patients will not wear the monobloc OA for 1 week (washout phase). Three months later - T2 (6 weeks of 'active' treatment), all the previous measurements will be conducted again.
  Interventions: Device: twinblock oral appliance
- oral appliance 1 (Experimental): Patients in treatment arm/group A will have a customized monobloc OA constructed for them individually. They will undergo an appliance acclimatization period of 4-5 weeks. Three months after baseline assessments - T1 (6 weeks of 'active' treatment), physiological measurements will be evaluated, clinical oral examinations conducted, quality of life and compliance assessed. Following this, a customized twin-bloc OA will be constructed for subjects individually and they will acclimatize to it for 4-5 weeks (so that the mandible is protruded to the maximum position they feel comfortable with when the appliance is worn). Prior to the active treatment phase, patients will not wear the twin-bloc OA for 1 week (washout phase). Three months later - T2 (6 weeks of 'active' treatment), all the previous measurements will be conducted again.
  Interventions: Device: monobloc oral appliance

INTERVENTIONS:
Device: monobloc oral appliance — one piece oral appliance
  Arms: oral appliance 1
Device: twinblock oral appliance — two-piece oral appliance
  Arms: oral appliance 2

SUMMARY:
Obstructive sleep apnoea (OSA) is a serious and common disorder affecting one in twenty-five men and one in fifty women over the age of 30. This breathing abnormality occurs during sleep and is characterised by snoring and episodes of sleep disturbances. The symptoms of untreated OSA (e.g. excessive daytime sleepiness), can result in significant reductions in the patients' quality of life. The key treatment modalities today include Continuous Positive Air Pressure (CPAP), surgery and the use of oral appliances (OAs). Increasingly, OAs have been advocated in the treatment of the symptoms of OSA since they offer a non-invasive form of treatment and also because patients often prefer this treatment to other treatment modalities. There is increasing evidence to support the effectiveness of OAs in the management of OSA, at least as a short term measure. What is still unclear is which types of OA are most effective and whether OAs are effective in the long term management of OSA. This randomized clinical trial aims to evaluate two differently designed OAs in terms of their effect on patients' quality of life and on the physiological symptoms of OSA (apnoea/hypopnoea index AHI). Around 45 patients with OSA will be recruited from a pool of patients referred to the dental hospital for treatment from the medical faculty. The treatment with OAs will commence after randomization to two treatment groups; follow-up examinations will take place over a period of 12 months. The results of this study will help inform practitioners and patients of the feasibility of using OAs in the long term management of OSA and help determine the most appropriate type of OAs for the management of OSA and improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* AHI ≥ 10-30/h, and those who do not tolerate CPAP or refused CPAP if AHI >30
* A score of > 10 on the Epworth Sleepiness Scale
* Body Mass Index <35kg/m
* Those who are competent to give written informed consent
* have adequate dental anchoring structures (<10 periodontally healthy teeth per arch)

Exclusion Criteria:

* Previous surgery to upper respiratory airway
* Concurrent unstable cardiovascular disease, neurological, mental or psychiatric disorders
* Recent major surgery in the last 6 months
* Pregnancy
* Epilepsy
* temporomandibular joint (TMJ) disfunction (pain during mandibular advancement or limitation of mouth opening)
* untreated dental decay

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 months
  Quality of life scores collected by the Sleep Apnoea Quality of Life Index questionnaire.
  The minimum important clinical difference (MICD) for this index is a change in score of 1. A mean change of at least 1 in the SAQLI scores (SD=1.1) between the two groups (treated two types of oral appliances) is expected.

SECONDARY OUTCOMES:
objective OSA markers | 6 months
  Physiological variables measured during polysomnography, such as apnea-hypopnea index (AHI).
  Complete response: Resolution of symptoms and improvement of objective variables Partial response: more than 50% reduction in AHI but AHI's remaining above 5/h Failure: ongoing clinincal symptoms and/or less than 50% reduction in AHI

CONTACTS AND LOCATIONS:
Overall Officials: Colman McGrath, Professor, Principal Investigator — Faculty of Dentistry, HKU
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, Hong Kong